CLINICAL TRIAL: NCT04383054
Title: Do Physical Activity (PA) Interventions Increase Acute Medical Inpatients Self-reported Physical Activity Levels (PAL): A Feasibility Study
Brief Title: Do PA Interventions Increase Acute Medical Inpatients PA Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19AM006
Record Dates: First submitted 2020-03-02; First posted 2020-05-11 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Physical Activity; Moving Medicine; Acute Medical Unit
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long PA intervention group (Experimental): The long PA intervention will be a MI (motivational interview) exploring the participant's knowledge and concerns about PA. An MI involves a semi-structured discussion between an investigator and the participant. The MI initially explores the participant's knowledge of the benefits of PA and their concerns about PA. The MI will then explore the participant's confidence in increasing their PAL, help the participant come up with a plan to increase their PAL and finally the participant will be signposted to further support and local opportunities for PA. The investigator will use a Moving Medicine 'more minutes' conversation tool of a chronic health condition that the patient has to facilitate every MI. Where possible the investigator will discuss the chronic condition that most relates to the participant's current admission to hospital. For patients with no health conditions the primary prevention section will be used.
  Interventions: Behavioral: 'More minutes' conversation (Moving medicine)
- Short PA intervention group (Active Comparator): The short PA intervention will involve a short (1 min) discussion between an investigator and a participant. A Moving Medicine 'one minute' intervention appropriate to the participant's health conditions will be used to guide every short intervention. The short intervention will firstly involve the investigator asking whether the participant knew that doing PA was beneficial for their health. The investigator would then explain to be more PA they could try to build more PA into their daily routine and that this was often enough to meet the current PA recommendations. The investigator will also offer the participant a patient information sheet about PA.
  Interventions: Behavioral: 'one minute' conversation (Moving medicine)

INTERVENTIONS:
Behavioral: 'More minutes' conversation (Moving medicine) — For the interventions in this study we have chosen to use the Moving Medicine conversation tools because they are an evidence-based PA intervention tool. The Moving Medicine 'more minutes' conversation tool initially involves the investigator exploring the participant's understanding of PA. Improving patients' knowledge of the benefits of PA may empower them to increase their PAL because knowledge of the benefits of PA may motivate patients to increase their PAL. The division of the Moving Medicine conversation tools into chronic health conditions is important because it will allow the investigator to explore topics relating to PA which are specific to the participant's own medical co-morbidities. For example, in a patient with known ischaemic heart disease the investigator could discuss how PA helps to prevent the risk of further heart attacks and the development of heart failure (Moving Medicine).
  Arms: Long PA intervention group
Behavioral: 'one minute' conversation (Moving medicine) — For the interventions in this study we have chosen to use the Moving Medicine conversation tools because they are an evidence-based PA intervention tool. The Moving Medicine 'more minutes' conversation tool initially involves the investigator exploring the participant's understanding of PA. Improving patients' knowledge of the benefits of PA may empower them to increase their PAL because knowledge of the benefits of PA may motivate patients to increase their PAL. The division of the Moving Medicine conversation tools into chronic health conditions is important because it will allow the investigator to explore topics relating to PA which are specific to the participant's own medical co-morbidities. For example, in a patient with known ischaemic heart disease the investigator could discuss how PA helps to prevent the risk of further heart attacks and the development of heart failure (Moving Medicine).
  Arms: Short PA intervention group

SUMMARY:
Physical activity (PA) can help treat and prevent many physical and mental health conditions. However, many of the United Kingdom population do not meet the Department of Health's PA recommendations which is contributing to the high chronic disease burden in the UK population. Many patients who are admitted to acute medical wards have at least one co- morbidity. Inpatients on acute hospital wards do not routinely receive PA advice from healthcare staff. The investigators believe that patients could be encouraged to increase their PA level (PAL) during an admission to hospital.

DETAILED DESCRIPTION:
The investigators have undertaken two previous qualitative studies that proceed this work. The first study found that patients were open to discussing PA during admission to an acute medical unit (AMU). In the second study patients thought motivational interviews focused on PA helped them increase their PAL. Although patients have reported that motivational interviews were beneficial in helping them increase their PA, this has so far not been assessed quantitatively.

The investigators plan to recruit 50-100 patients and randomise them into two groups. One group will receive a short PA intervention and the other a long intervention. The investigators will use the moving medicine online resource to structure both PA intervention. The 'one minute' conversation will be used for the short PA intervention and the 'more minutes' conversation for the long PA intervention. The investigators will measure the PAL of both groups at baseline and at two follow-up points (4 weeks and 12 weeks). The Global Physical Activity Questionnaire will be used to assess participants self-reported PAL. The data collected will be used to describe participants baseline PAL and the treatment effect of the two PA interventions. The investigators will also calculate estimated recruitment and retention rates. The results of this feasibility study will be used to plan a similarly designed powered randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* Patients equal or greater than 18 years of age.
* Patients identified by ward staff as being about to be discharged from hospital over the coming day(s).
* Patients identified by ward staff as being able to walk 10m on flat ground, with or without a walking aid.

Exclusion Criteria:

* Patients who do not understand verbal and written English.
* Patients who currently meet the Department of Health's current aerobic physical activity recommendations as assessed by the GPAQ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Participant's self reported Metabolic Equivalents (METs) at 4 weeks assessed using the Global Physical Activity Questionnaire. | 4 weeks
  The primary outcome is the participant's physical activity level (PAL) at the 4 week follow-up point. The investigators will use the Global Physical Activity Questionnaire (GPAQ) to assess participant's PAL. The GPAQ will be analysed using the GPAQ analysis guide to provide a result in Metabolic Equivalents (METs). MET is the ratio of a person's working metabolic rate relative to the resting metabolic rate and is commonly used to express the intensity of physical activities. One MET is defined as the energy cost of sitting quietly. MET is therefore a linear scale of physical activity (PA) from 0 upwards with no maximum value. The higher the MET the more PA a person is doing. The Department of Health advise adults to do a combination of moderate to vigorous PA totalling 150 minutes of moderate PA or 75 minutes of vigorous PA a week (or a combination of both). The approximate MET equivalent of 150 minutes of moderate intensity PA is 600 METs

SECONDARY OUTCOMES:
Participant's self reported Metabolic Equivalents (METs) at 12 weeks assessed using the Global Physical Activity Questionnaire | 12 weeks
  The primary outcome is the participant's physical activity level (PAL) at the 12 week follow-up point. The investigators will use the Global Physical Activity Questionnaire (GPAQ) to assess participant's PAL.The GPAQ will be analysed using the GPAQ analysis guide to provide a result in Metabolic Equivalents (METs). MET is the ratio of a person's working metabolic rate relative to the resting metabolic rate and is commonly used to express the intensity of physical activities. One MET is defined as the energy cost of sitting quietly. MET is therefore a linear scale of physical activity (PA) from 0 upwards with no maximum value. The higher the MET the more PA a person is doing. The Department of Health advise adults to do a combination of moderate to vigorous PA totalling 150 minutes of moderate PA or 75 minutes of vigorous PA a week (or a combination of both). The approximate MET equivalent of 150 minutes of moderate intensity PA is 600 METs
physical activity level at baseline | baseline
  The primary outcome is the participant's physical activity level at baseline. The investigators will use the Global Physical Activity Questionnaire (GPAQ) to assess participant's physical activity level. The GPAQ will be analysed using the GPAQ analysis guide to provides a result in a METs.
recruitment rate | 1-2 months
  the number of days taken to recruit 50 participants
retention rate | 3 months
  the number of participants who complete the 4 and 12 week follow-up points

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Medical Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No